CLINICAL TRIAL: NCT06348134
Title: Assessing the Efficacy and Safety of Optimal Neoadjuvant to Adjuvant Anti-HER2- Based Therapy in Nigerian Women With HER2+ Breast Cancer
Brief Title: Assessing the Efficacy and Safety of Anti-HER2 Therapy in Nigerian Women With HER2+ Breast Cancer Before and After Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0502
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-02

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; HER2-positive Breast Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; pertuzumab; Docetaxel; Tamoxifen; Letrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: All Participants (Experimental): All participants will receive a combination of:
  * docetaxel (starting dose - 75 mg/m2), increasing to 100mg/m2 by cycle 2 (if tolerated) for 4-6 cycles (for a total of 18 weeks). Docetaxel will be give as an injection.
  * trastuzumab and pertuzumab (loading dose of 1200 mg of pertuzumab and 600 mg trastuzumab) for 52 weeks followed by 600 mg pertuzumab and 600 mg trastuzumab every 3 weeks for 15 cycles (for a total of 52 weeks). These two drugs will be given as subcutaneous injections under the skin.
  Interventions: Drug: Trastuzumab emtansine; Drug: Pertuzumab Injection; Drug: Docetaxel
- Phase 2 - Operable (participants who are able to have surgery) (Experimental): Participants in this group will have breast cancer that shows a complete or incomplete response (as assessed by ultrasound) to the study drug combination given in phase 1 of study. Based on how their breast cancer responds to the phase 1 study drugs, participants in this group will:
  - undergo surgery and will continue to receive pertuzumab (600 mg) and trastuzumab (600 mg) for 36 weeks. Participants may also receive hormone therapy (as recommended by study doctor) based on status of breast cancer. This drug will be given as an injection under the skin.
  Some participants in this group may also receive tamoxifen (as an oral tablet; 20 mg daily for 10 years after surgery), letrozole (as an oral tablet 2.5 mg daily for 10 years after surgery) and/or goserelin (hormone injection 10.8 mg every 1-3 months) based on their human epidermal growth factor receptor 2 (HER2) status as assessed by the treating doctor.
  Interventions: Drug: Trastuzumab emtansine; Drug: Pertuzumab Injection; Drug: Docetaxel; Drug: Tamoxifen; Drug: Letrozole; Drug: Goserelin
- Phase 2 - Inoperable (participants who are not able to have surgery) (Experimental): Participants in this group will have breast cancer that shows a partial response (as assessed by ultrasound) to the study drugs given in phase 1 or their breast cancer stayed the same or got worse after receiving study drugs during phase 1. Based on how their breast cancer responds to the phase 1 study drug regimen, participants in this group will receive trastuzumab emtansine (intravenously) plus standard chemotherapy as recommended by their doctor.
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine — A chemotherapy drug.
  Other Names: Kadcyla; T-DMI
Drug: Pertuzumab Injection — A prescription medicine that is approved for use in combination with trastuzumab and docetaxel in people who have HER2-positive breast cancer that has spread to different parts of the body (metastatic) and who have not received anti-HER2 therapy or chemotherapy for metastatic breast cancer.
  Other Names: Perjeta
  Arms: Phase 1: All Participants; Phase 2 - Operable (participants who are able to have surgery)
Drug: Docetaxel — A chemotherapy drug.
  Other Names: Taxotere; Docefrez
  Arms: Phase 1: All Participants; Phase 2 - Operable (participants who are able to have surgery)
Drug: Tamoxifen — A medication used to treat breast cancer.
  Other Names: Soltamox
  Arms: Phase 2 - Operable (participants who are able to have surgery)
Drug: Letrozole — A medication used to treat breast cancer.
  Arms: Phase 2 - Operable (participants who are able to have surgery)
Drug: Goserelin — A hormone therapy drug.
  Other Names: Zoladex
  Arms: Phase 2 - Operable (participants who are able to have surgery)

SUMMARY:
Doctors leading this study would like to learn about providing cancer treatment/therapies to Nigerian women with breast cancer based on their human epidermal growth factor receptor 2 (HER2) status. This study will focus on the efficacy and safety of anti-HER2 cancer treatment before and after surgery.

DETAILED DESCRIPTION:
Doctors leading this study would like to learn about providing cancer treatment/therapies to Nigerian women with breast cancer based on their human epidermal growth factor receptor 2 (HER2) status. This study will focus on the efficacy and safety of anti-HER2 cancer treatment before and after surgery. Participants with HER2-positive breast cancer will receive a combination of trastuzumab with pertuzumab (PHESGO) plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any screening procedures

1. Women ages of 18 to 70 years old
2. Biopsy-accessible breast tumor of significant size for core needle biopsy /ultrasound measurable (≥ 2cm)
3. Measurable breast tumour using ultrasonography (≥ 2cm)
4. Patients with histologically confirmed carcinoma of the female breast with positive HER2 status
5. Clinical stages 2A -3C. (AJCC 2009)
6. Chemotherapy-naïve patients (for this malignancy)
7. Performance status: Eastern Cooperative Oncology Group performance status 0-3
8. Non-pregnant and not nursing. Women of childbearing potential must take the pregnancy test and must commit to receive hormone therapy with Zoladex (goserelin) for two years starting from the commencement of the study medications
9. Required Initial Laboratory Data. Adequate hematologic, renal and hepatic function, as defined by each of the following:

1. Granulocyte ≥ 1,500/mL 2. Platelet count ≥ 100,000/mL 3. Absolute neutrophil count ≥ l500/mL 4. Hemoglobin 10g/dL 5. Bilirubin ≤ 1.5 x upper limit of normal 6. serum glutamic-oxaloacetic transaminase (SGOT) and Serum glutamic pyruvic transaminase (SGPT) < 2.5 x upper limit of normal for patients without liver metastases 7. Creatinine within institutional normal limits or glomerular filtration rate ≥ 30 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration equation (see http://mdrd.com/ for calculator) 8. Echocardiogram: Baseline left ventricular ejection fraction of ≥ 55%

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Pregnant or lactating women. Women of childbearing potential not using a reliable and appropriate contraceptive method. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Patients will agree to continue the use of acceptable form of contraception for 7 months from the date of last drug administration (Herceptin).
2. Patients with distant metastasis
3. Serious, uncontrolled, concurrent infection(s).
4. Patients who have received more than 4 weeks of tamoxifen therapy for this malignancy. Patient who have received tamoxifen or raloxifene for purposes of chemoprevention (e.g. Breast Cancer Prevention Trial or for other past indications (including previous breast cancer) are eligible. Tamoxifen or raloxifene therapy will be discontinued at least one month before the patient is enrolled on this study.
5. Treatment for other carcinomas within the last 5 years, except non-melanoma skin cancer and treated cervical carcinoma in-situ (CCIS)
6. Participation in any investigational drug study within 4 weeks preceding the start of study treatment
7. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation including but not limited to chronic or active infection, HIV-positive patient, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled Diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Unwillingness to participate or inability to comply with the protocol for the duration of the study
9. Patients with human epidermal growth factor receptor 2 (HER2-negative) disease
10. History of documented heart failure or systolic dysfunction (LVEF < 50%), High-risk uncontrolled arrhythmias ie, atrial tachycardia with a heart rate > 100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade Atrioventricular (AV)-block (second degree AV-block Type 2 [Mobitz 2] or third degree AV-block),
11. Angina pectoris requiring anti-anginal medication,
12. Clinically significant valvular heart disease
13. Poorly controlled hypertension (eg, systolic > 180 mm Hg or diastolic > 100 mm Hg)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer study.
Enrollment: 74 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2034-07-01 (Estimated); Study Completion 2036-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | 10 years
  Pathological complete response of giving three-weekly docetaxel + subcutaneous trastuzumab and Pertuzumab with Tamoxifen/Letrozole added ) to Nigerian women with Human epidermal growth factor receptor 2 (HER2-positive) breast cancer as assessed by the absence of invasive neoplastic cells at microscopic examination of the primary tumor and lymph nodes at surgery.

SECONDARY OUTCOMES:
Reported Adverse Events and clinical/medical records of participants | 10 years
  Reported adverse events among participants receiving three-weekly docetaxel + subcutaneous trastuzumab and Pertuzumab with Tamoxifen/Letrozole added ) to Nigerian women with Human epidermal growth factor receptor 2 (HER2-positive) breast cancer as assessed by the incidence and severity of adverse events and serious adverse drug reactions including clinical laboratory values, vital signs, electrocardiogram and dose interruptions. Adverse events will be defined by the Common Terminology Criteria for Adverse Events (CTCAE Grade 4)
Percentage of participants who are suitable for breast-conserving surgery | 10 years
  To determine suitability of patients for breast conserving surgery after neoadjuvant treatment with docetaxel and PHESGO as assessed by the percentage of patients with breast conservative surgery following neoadjuvant therapy.
Event-free survival duration reported among participants | 10 years
  Event-free responses defined as time from first dose of study drug treatment to progression or death due to any cause, as assessed by investigators.
Quality of life reported among study participants | 10 years
  Quality of life (QoL) will be assessed by various domains of QoL over time and the changes from baseline using a QoL instrument (a global/breast module) validated by the European Organization for Research and Treatment of Cancer (EORTC). QLQ-C30 version 3.0 and Breast Cancer Module QLQ-BR23 low scores on scale of 0-4 indicates better financial wellbeing
Genetic and epigenetic factors associated with breast cancer in Nigeria | 10 years
  To assess the genetic and epigenetic factors associated with breast cancer in Nigeria asa assessed by correlative study of molecular markers and tumor subtypes/tumor biology with patient's characteristics, response or resistance to treatment and participants' outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo Olopade, Principal Investigator — University of Chicago
Locations (5):
- University of Chicago, Chicago, Illinois, United States
- Nigeria (4):
  - Lagos State University Teaching Hospital, Ikeja, Lagos
  - Lagos University Teaching Hospital, Yaba, Lagos
  - Obafemi Awolowo University Teaching Hospitals Complex (OAUTHC), Ile-Ife, Osun State
  - University of Ibadan Hospital, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF